CLINICAL TRIAL: NCT03024255
Title: A Multicenter, Randomized, Double-Blinded, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of 3 Concentrations of Topically Applied BBI-4000 (Sofpironium Bromide) Gel in Subjects With Axillary Hyperhidrosis
Brief Title: A Confirmatory Safety and Efficacy Study of BBI-4000 in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI-4000-CL-203
Record Dates: First submitted 2017-01-06; First posted 2017-01-18 (Estimated); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Hyperhidrosis
Keywords: sweat gland disease; sweating; underarm
MeSH Terms: conditions — Hyperhidrosis; Sweat Gland Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BBI-4000 gel, 5% (Experimental): BBI-4000 gel, 5% applied once to each axilla daily
  Interventions: Drug: BBI-4000 gel, 5%
- BBI-4000 gel, 10% (Experimental): BBI-4000 gel, 10% applied once to each axilla daily
  Interventions: Drug: BBI-4000 gel, 10%
- BBI-4000 gel, 15% (Experimental): BBI-4000 gel, 15% applied once to each axilla daily
  Interventions: Drug: BBI-4000 gel, 15%
- Vehicle (Placebo Comparator): Placebo, applied once to each axilla daily
  Interventions: Drug: Vehicle (Placebo)

INTERVENTIONS:
Drug: BBI-4000 gel, 5% — BBI-4000 gel, 5% applied once to each axilla daily
  Other Names: BBI-4000 Low Concentration
  Arms: BBI-4000 gel, 5%
Drug: BBI-4000 gel, 10% — BBI-4000 gel, 10% applied once to each axilla daily
  Other Names: BBI-4000 Medium Concentration
  Arms: BBI-4000 gel, 10%
Drug: BBI-4000 gel, 15% — BBI-4000 gel, 15% applied once to each axilla daily
  Other Names: BBI-4000 High Concentration
  Arms: BBI-4000 gel, 15%
Drug: Vehicle (Placebo) — Placebo, applied once to each axilla daily
  Other Names: Control
  Arms: Vehicle

SUMMARY:
This study is being conducted to assess the safety and efficacy of 3 concentrations of BBI-4000 and vehicle (4 treatment arms), applied for the treatment of axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a Multicenter, Randomized, Double Blind, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of 3 concentrations of Topically Applied BBI-4000 in Subjects with Axillary Hyperhidrosis.

Safety will be assessed through collection of vital signs, adverse events, local skin responses, hematology, serum chemistry laboratory testing and urinalysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥ 18 years of age.
* Diagnosis of primary axillary hyperhidrosis that meets the following criteria: (a) symptoms of hyperhydrosis for at least 6 months' duration, (b) HDSM-Ax of 3 - 4, (c) HDSS of 3 or 4 and (d) a minimum GSP of 50 mg is each axilla with a combined total of at least 150 mg.
* The ability to understand and follow all study-related procedures including study drug administration.
* Sexually active female of childbearing potential (FOCBP)* must agree to periodic pregnancy testing and use a medically acceptable method of contraception while receiving protocol-assigned product.

Exclusion Criteria:

* In the Investigators opinion, any skin or subcutaneous tissue conditions of the axilla(s).
* Prior use of any prohibited medication(s) or procedure(s) within the specified timeframe for the treatment of axillary hyperhidrosis.
* Anticholinergic agents used to treat conditions such as, but not limited to, hyperhidrosis, asthma, incontinence, gastrointestinal cramps, and muscular spasms by any route of administration.
* Use of potent inhibitors of cytochrome P450 CYP3A and CYP2D6.
* Use of any cholinergic drug (e.g. bethanechol) within 30 days.
* Known cause of hyperhidrosis or known history of a condition that may cause hyperhidrosis (i.e., hyperhidrosis secondary to any known cause such hyperthyroidism, diabetes mellitus, medications, etc.).
* Subjects with unstable diabetes mellitus or thyroid disease, history of renal or hepatic impairment, malignancy glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, BPH, neurological or psychiatric conditions, Sjögren's or Sicca syndrome, or cardiac abnormalities that may alter or exacerbate sweat production by the use of anticholinergics in the investigator's opinion.
* Subjects with known hypersensitivity to glycopyrrolate, anticholinergics, or any of the components of the topical formulation.
* Subject is pregnant, lactating or is planning to become pregnant during the study.
* History or presence of supraventricular tachycardia, ventricular arrhythmias, atrial fibrillation or atrial flutter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD PhD, Study Director — Botanix Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vehicle: Vehicle (Placebo), applied once to each axilla daily
Period: Overall Study
Arm/Group | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Vehicle
Started | 57 | 57 | 56 | 57
Completed | 50 | 49 | 45 | 52
Not Completed | 7 | 8 | 11 | 5
Not completed — Adverse Event | 1 | 4 | 8 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Protocol Noncompliance | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population includes all subjects randomized in the study who received study drug at least once. Treatment group assignment was based on the treatment actually received. Two participants were randomized to BBI-4000 gel, 15% but were not dispensed the medication.
Groups:
- Vehicle: Vehicle (Placebo), administered to each axilla once daily
- BBI-4000 Gel, 5%: BBI-4000 gel, 5% administered to each axilla once daily
- BBI-4000 Gel, 10%: BBI-4000 gel, 10% administered to each axilla once daily
- BBI-4000 Gel, 15%: BBI-4000 gel, 15% administered to each axilla once daily
- Total: Total of all reporting groups
Arm/Group | Vehicle | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15% | Total
Number analyzed (Participants) | 57 | 57 | 57 | 54 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (8.62) | 30.8 (10.22) | 33.7 (11.29) | 30.7 (9.24) | 31.3 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 22 | 25 | 102
  Male | 27 | 32 | 35 | 29 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 8 | 12 | 15 | 48
  Not Hispanic or Latino | 44 | 49 | 45 | 39 | 177
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Subjects reporting more than one race were originally included in all relevant race categories. Percentages added up to >100%. For this table, subjects reporting more than one race were categorized only into "More Than One Race".
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
    Asian | 1 | 3 | 3 | 2 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 10 | 4 | 9 | 10 | 33
    White | 41 | 47 | 44 | 42 | 174
    More than one race | 3 | 2 | 1 | 0 | 6
    Unknown or Not Reported | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change of Hyperhidrosis Disease Severity Measure-Axillary (HDSM-Ax) Score From Baseline to End of Therapy
Description: 11 question evaluation tool to assess the effect of BBI-4000 gel, 5%, 10% and 15 % on hyperhidrosis disease severity measures in subjects with axillary hyperhidrosis. Two questions measured the frequency (since yesterday) of underarm sweating outcomes. The range of responses included increasing frequency scale: None of the time (0); A little of the time (1); Some of the time (2); Most of the time (3); All of the time (4). The next seven questions measured the severity of underarm sweating outcomes. Range in increasing severity: I did not experience this (0); Mild (1); Moderate (2); Severe (3); Very Severe (4). The last two questions measured the need to change or clean from underarm sweating. Range in increasing degree of need: Not at all (0); Slight (1); Moderate (2); Strong (3); Very Strong (4).
  The mean was derived by taking the total score and dividing by the number of questions answered. A negative LSM reflects a reduction, decrease or measured improvement in HDSM-Ax
Time Frame: overall ~6 Weeks, as listed in description includes: Baseline-Visit 1, Visit 4 and End of Therapy Visit - Days 41, 42, 43.
Population: mITT Population
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Groups:
- Vehicle: Vehicle (Placebo), applied to each axilla once daily
- BBI-4000 Gel, 5%: BBBI-4000 Sofpironium Bromide Gel, 5% applied to each axilla once daily
- BBI-4000 Gel, 10%: BBBI-4000 Sofpironium Bromide Gel, 10% applied to each axilla once daily
- BBI-4000 Gel, 15%: BBBI-4000 Sofpironium Bromide Gel, 15% applied to each axilla once daily
Arm/Group | Vehicle | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15%
Number analyzed (Participants) | 53 | 52 | 50 | 47
score on a scale | -1.30 (0.136) | -2.02 (0.135) | -2.09 (0.137) | -2.10 (0.143)

2. Primary Outcome: Number (%) of Subjects Reporting at Least One Treatment Emergent Adverse Event by Severity
Description: Subjects reporting more than one adverse event are counted only once using the highest severity.
Time Frame: Treatment initiation through end of treatment (~42 days) and subsequent safety f/u (~14 days following end of treatment)
Population: Number (%) of Subjects Reporting at Least One: TEAE n(%), Safety Population: Vehicle (N=57), BBI-4000 5% (N=57), BBI-4000 10% (N=57), BBI-4000 15% (N=54)
Measure: Count of Participants; unit: Participants
Groups:
- BBI-4000 Gel, 10%: BBI-4000 Sofpironium Bromide Gel, 10% applied to each axilla once daily
- BBI-4000 Gel, 15%: BBI-4000 Sofpironium Bromide Gel, 15% applied to each axilla once daily
Arm/Group | Vehicle | BBI-4000 Gel, 5% | BBI-4000 Gel, 10% | BBI-4000 Gel, 15%
Number analyzed (Participants) | 9 | 17 | 19 | 28
Participants
  Mild | 7 | 7 | 10 | 11
  Moderate | 2 | 8 | 7 | 13
  Severe | 0 | 2 | 2 | 4

3. Secondary Outcome: Average Gravimetrically Measured Sweat Production (GSP) Observed by Visit, Per Protocol Population
Description: Measured weight of the amount of sweat produced by Visit Method of calculating average for Baseline, End of Therapy, and End of Therapy Imputed.
  Baseline GSP was defined as the mean of any available Visit 2, Visit 3, and Visit 4 values (occurring Days -21 to -7 relative to Day 1 Baseline) End of Therapy is defined as the mean of any available Day 41, Day 42, and Day 43 values.
Time Frame: Visit 2, 3, and 4 timepoints were reported Days -21 to -7, relative to Visit 5/ Day 1/Baseline, Days 8, 15, 22, 29, 36, 41, 42, 43, and 57
Population: Overall number of participants analyzed includes those who were compliant with the protocol. Compliance with the protocol per visit at Visits 2-4 (Days -21 to -7), Baseline Visit (Day 1), and Days 8, 15, 22, 29, 36, 41, 42, 43, and 57, affected the number of participants analyzed at these timepoints.
Measure: Mean (Standard Deviation); unit: Combined Axilla GSP (mg)
Units Other Than Participants: Both axilla combined total
Groups:
- Vehicle: Vehicle (Placebo) Applied to each axilla once daily
- BBI-4000 Gel 5%: BBI-4000 Sofpironium Bromide Gel 5% applied to each axilla once daily
- BBI-4000 Gel 10%: BBI-4000 Sofipironium Bromide Gel 10% applied to each axilla once daily
- BBI-4000 Gel 15%: BBI-4000 Sofpironium Bromide Gel 15% applied to each axilla once daily
Arm/Group | Vehicle | BBI-4000 Gel 5% | BBI-4000 Gel 10% | BBI-4000 Gel 15%
Number analyzed (Participants) | 50 | 49 | 47 | 44
Number analyzed (Both axilla combined total) | 100 | 98 | 94 | 88
Combined Axilla GSP (mg)
  Baseline | 259.53 (141.738) | 282.41 (201.920) | 281.63 (211.542) | 316.39 (201.478)
  Day 8: number analyzed (Participants) | 48 | 47 | 45 | 44
  Day 8: number analyzed (Both axilla combined total) | 96 | 94 | 90 | 88
  Day 8 | 137.36 (144.104) | 124.94 (199.072) | 113.77 (119.233) | 118.49 (129.393)
  Day 15: number analyzed (Participants) | 48 | 48 | 45 | 41
  Day 15: number analyzed (Both axilla combined total) | 96 | 98 | 90 | 82
  Day 15 | 131.50 (100.171) | 114.24 (175.195) | 114.07 (169.784) | 106.68 (121.225)
  Day 22: number analyzed (Participants) | 49 | 49 | 47 | 44
  Day 22: number analyzed (Both axilla combined total) | 98 | 98 | 94 | 88
  Day 22 | 141.10 (153.886) | 102.43 (213.006) | 112.34 (128.033) | 90.48 (98.380)
  Day 29: number analyzed (Participants) | 50 | 49 | 46 | 41
  Day 29: number analyzed (Both axilla combined total) | 100 | 98 | 92 | 82
  Day 29 | 114.12 (91.999) | 106.06 (180.981) | 168.13 (230.825) | 117.60 (135.284)
  Day 36: number analyzed (Participants) | 49 | 46 | 46 | 44
  Day 36: number analyzed (Both axilla combined total) | 98 | 92 | 92 | 88
  Day 36 | 142.87 (156.561) | 105.16 (200.641) | 124.33 (147.519) | 126.44 (231.723)
  Day 41 | 116.61 (132.620) | 119.00 (195.636) | 117.85 (141.070) | 93.21 (131.063)
  Day 42 | 110.96 (161.590) | 95.09 (157.573) | 111.98 (140.927) | 88.62 (103.408)
  Day 43 | 159.13 (157.113) | 139.65 (291.857) | 105.03 (108.026) | 117.34 (159.217)
  Day 57 | 163.43 (193.565) | 112.09 (181.185) | 177.62 (242.634) | 135.76 (165.620)

ADVERSE EVENTS:
Time Frame: Treatment-Emergent Adverse Events (TEAEs) were collected from during investigational treatment Days 1 to 42. A safety follow-up assessment including of TEAEs was also performed ~14 days post end of treatment. A total of 225 subjects were included in the Safety population (54 subjects in the 15% group; and 57 subjects each in the 10%, 5%, and vehicle groups).
Description: Treatment-Emergent Adverse Events by System Organ Class and Preferred Term (Safety Population)
Groups:
- Vehicle: Vehicle (Placebo), applied to each axilla, once daily
- BBI-4000 Sofpironium Bromide Gel 5%: BBI-4000 Sofpironium Bromide Gel 5%, applied to each axilla, once daily
- BBI-4000 Sofpironium Bromide Gel 10%: BBI-4000 Sofpironium Bromide Gel 10%, applied to each axilla, once daily
- BBI-4000 Sofpironium Bromide Gel 15%: BBI-4000 Sofpironium Bromide Gel 15%, applied to each axilla, once daily
Arm/Group | Vehicle | BBI-4000 Sofpironium Bromide Gel 5% | BBI-4000 Sofpironium Bromide Gel 10% | BBI-4000 Sofpironium Bromide Gel 15%
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57 | 0/57 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/57 | 1/57 | 0/57 | 0/54
Other Adverse Events (participants affected / at risk) | 9/57 | 17/57 | 19/57 | 28/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=57) | BBI-4000 Sofpironium Bromide Gel 5% (N=57) | BBI-4000 Sofpironium Bromide Gel 10% (N=57) | BBI-4000 Sofpironium Bromide Gel 15% (N=54)
Staphylococcal osteomyelitis / T8-T9 osteomyelitis/discitis with biopsy positive for streptococcus a (Infections and infestations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=57) | BBI-4000 Sofpironium Bromide Gel 5% (N=57) | BBI-4000 Sofpironium Bromide Gel 10% (N=57) | BBI-4000 Sofpironium Bromide Gel 15% (N=54)
Dry Mouth (Gastrointestinal disorders) | 1 | 9 | 10 | 12
Vision Blurred (Eye disorders) | 0 | 2 | 6 | 5
Application Site Pain (General disorders) | 0 | 1 | 3 | 5
Application Site Pruritus (General disorders) | 0 | 0 | 3 | 3
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 2 | 4
Dry eye (Eye disorders) | 0 | 2 | 2 | 1
Application site dermatitis (General disorders) | 0 | 3 | 1 | 0
Application site erythema (General disorders) | 0 | 1 | 1 | 2
Application site rash (General disorders) | 0 | 1 | 0 | 2
Application site folliculitis (General disorders) | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Application site irritation (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Application site dryness (General disorders) | 0 | 0 | 0 | 1
Application site erosion (General disorders) | 0 | 0 | 0 | 1
Application site exfoliation (General disorders) | 0 | 0 | 0 | 1
Application site odour (General disorders) | 0 | 0 | 1 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Mydriasis (Eye disorders) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0
Heliobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0
Osteomyelitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement terms prioritized a multi-center publication at the study end. Should such a publication not be completed, an investigator right to individually publish results of his/her study (limited to his/her site data) was included, if for purely scientific or educational purposes; not for any commercial purposes. PI(s) were to submit draft materials to the Sponsor 60 days prior to Investigator release of individual abstract or manuscript. Additional disclosure restrictions and terms applied .

DOCUMENTS (2):
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03024255/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT03024255/SAP_001.pdf